CLINICAL TRIAL: NCT03624530
Title: Effect of Prophylactic Tyrosine Kinase Inhibitor Therapy Post-transplants on Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia Undergoing Allo-HSCT With Minimal Residual Disease Positive Pre-transplants
Brief Title: Effect of Prophylactic TKI Therapy Post-transplants on Ph+ ALL Undergoing Allo-HSCT With MRD Positive Pre-transplants
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Zhujiang Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKI post-HSCT- MRD+Ph+ALL-2018
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Philadelphia Chromosome Positive Acute Lymphocytic Leukemia; Tyrosine Kinase Inhibitor; Minimal Residual Disease; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Neoplasm, Residual | interventions — Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic TKI Therapy (Experimental): Treatment with prophylactic TKI will be initiated from day +30 to +60 post-transplants. TKI was selected according to the mutation results of ABL kinase region.
  Interventions: Drug: Tyrosine kinase inhibitor (TKIs)
- No TKI therapy (No Intervention): Prophylactic TKI will not be given.

INTERVENTIONS:
Drug: Tyrosine kinase inhibitor (TKIs) — TKI was selected according to the mutation results of ABL kinase region. Imatinib was initiated at a dose of 200mg/d, dasatinib at a dose of 50mg/d, and ponatinib at a dose of 30mg/d. Then increase the dosage of TKI gradually and increase to therapeutic dose within one month. The duration of TKI was 180 days.
  Arms: Prophylactic TKI Therapy

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) in early first complete remission improves the long-term outcomes for Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL). Relapse remains a major cause of treatment failure even after allo-HSCT. The prevention of relapse is essential for improving the outcome of Ph+ ALL. Our previous clinical trial (ID: NCT01883219) demonstrated that pre-emptive tyrosine kinase inhibitor (TKIs) administration based on minimal residual disease (MRD) and BCR-ABL mutation after allo-HSCT might reduce the incidence of relapses and improve survival for patients with Ph+ ALL. Moreover, our result suggested that Ph+ ALL with MRD positive pre-transplants had the higher rate of molecular biology relapse. In this study, we will evaluate the safety and efficacy of prophylactic TKI therapy post-transplants on Ph+ ALL undergoing allo-HSCT with MRD positive pre-transplants.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) in early first complete remission improves the long-term outcomes for Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL). Relapse remains a major cause of treatment failure even after allo-HSCT. Overall, patients experiencing relapse have a dismal prognosis despite salvage treatment with TKIs. The prevention of relapse is essential for improving the outcome of Ph+ ALL. Strategies to prevent relapse include tyrosine kinase inhibitor (TKIs) use, donor lymphocyte infusions (DLI), CAR-T and so on. At present, the utility of TKIs administration post-transplants is controversial. Our previous clinical trial (ID: NCT01883219) demonstrated that pre-emptive TKI administration based on minimal residual disease (MRD) and BCR-ABL mutation after allo-HSCT might reduce the incidence of relapses and improve survival for patients with Ph+ ALL. Moreover, we found that 58% Ph+ ALL with MRD positive pre-transplants would MRD positive post-transplants, whereas only 11.4% Ph+ ALL with MRD negative pre-transplants would MRD positive post-transplants, suggesting that Ph+ ALL with MRD positive pre-transplants had the higher rate of molecular biology relapse. In this study, we will evaluate the safety and efficacy of prophylactic TKI therapy post-transplants on Ph+ ALL undergoing allo-HSCT with MRD positive pre-transplants.

ELIGIBILITY:
Inclusion Criteria:

* Patient age of 14-65 years
* Ph+ ALL undergoing allo-HSCT with MRD positive pre-transplants
* Survival > 30 days post-transplants
* MRD negative on day +30 post-transplants

Exclusion Criteria:

* Ph+ ALL undergoing allo-HSCT with MRD negative pre-transplants
* Survival <30 days post-transplants
* MRD positive on day +30 post-transplants
* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 2 year
  the time from the date of transplantation to death or the last day of follow-up

SECONDARY OUTCOMES:
Relapse rate | 2 year
  the cumulative relapse rate of leukemia
Disease-free survival(DFS) | 2 year
  the time from the date of transplantation to relapse or death or the last day of follow-up
Adverse effects of TKI therapy | 2 year
  Number of participants with treatment-related adverse events and specific adverse effects including fluid retention , diarrhea, headache, nausea, rash, dyspnea, bleeding, fatigue, musculoskeletal pain, infection, vomiting, cough, abdominal pain and fever.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China